CLINICAL TRIAL: NCT00133809
Title: Islet Transplantation in Type 1 Diabetes Using the Edmonton Protocol of Steroid Free Immunosuppression
Brief Title: Islet Transplantation in Type 1 Diabetics Using the Edmonton Protocol of Steroid Free Immunosuppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Nicole Turgeon MD, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00041120; 10402 (Other: Other)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; Islet Transplantation; Immunology
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Islet Transplant (Experimental): All subjects who are found eligible and who can be matched to an appropriate donor will receive/have received an islet transplant
  Interventions: Drug: Transplantation of Human Islets

INTERVENTIONS:
Drug: Transplantation of Human Islets — Human islets, at least 9,000 islet equivalents per kilogram of body weight. Transplant involves surgical procedure

SUMMARY:
This trial will study the ability of islet transplantation to restore glycemic control and achieve insulin independence in type 1 diabetic subjects with life-threatening hypoglycemia and unawareness, or recurrent hyperglycemia with ketoacidosis.

DETAILED DESCRIPTION:
LAY SUMMARY:

More than 1 million North Americans have type 1 diabetes. Each year, approximately 30,000 new cases of type 1 diabetes are diagnosed in the United States. Type 1 diabetes destroys islets, a cluster of cells within the pancreas that produce insulin. Insulin is a hormone with many effects. However, the most important effect of insulin is to control the level of sugar in the blood. People with Type 1 diabetes no longer produce insulin and must take insulin injections to live. Despite steady improvements in the management of this disease, its victims remain at increased risk for stroke, heart attack, kidney failure, amputation, blindness, nerve damage and premature death. The life expectancy of a teenager is reduced by thirty years from the time of onset of the disease. Unfortunately, many type 1 diabetics cannot control their blood sugars in spite of very careful monitoring and the frequent injection of insulin. This group of patients is considered to have labile or "brittle" diabetes. These "brittle" diabetics can often have wide swings in their blood sugar levels that can be life threatening. Hypoglycemia, or low blood sugars, occurs when too much insulin is in the bloodstream. When this occurs, it is vital that patients eat or drink something right away that will increase their blood sugars. Many diabetics lose the ability to recognize when their blood sugars are getting dangerously low. These episodes of hypoglycemia can lead to coma, and possibly death, if not recognized and treated right away. Patients can also experience extreme increases in blood sugars, or hyperglycemia, as a result of emotional or physical stress. Hyperglycemia can result in dehydration, confusion, and a condition called ketoacidosis, which can lead to death. When this happens, insulin must be given as soon as possible.

Islet transplantation can restore the body's ability to make insulin and, in turn, restore normal blood sugar levels.

Since the 1960's, doctors and scientists have attempted to replace this islet function by performing whole organ pancreas transplantation. While the results of pancreas transplantation have improved dramatically in recent years, this approach has largely been limited to patients with kidney disease who have also needed a kidney transplant. This is because of the risks associated with the surgical procedure and the immunosuppressive drugs required to prevent rejection or the destruction of the transplanted pancreas by the body's immune system. Transplantation of a whole pancreas requires a major operation that is done through an incision in the abdomen. The patient must be under general anesthesia, or asleep, for the entire procedure. Recent clinical experience suggests that islet transplantation may be a useful approach to correct diabetes in humans.

Islet transplantation offers a direct approach to the treatment of type 1 diabetes. A large number of experimental studies carried out in many laboratories over the last decade have documented the beneficial effects of islet transplants in experimental animals. These experiments have confirmed both the efficiency and safety of islet transplantation.

The inability to isolate enough islets from a single pancreas has been one obstacle to successful islet transplantation. A certain number of islets must be isolated, or separated, from a single pancreas in order to use them for transplant. If this minimum number of islets is not obtained, then the islets do not effectively reverse diabetes. Progress in isolating the islets from a human pancreas has been dramatic in the last several years. Advances in equipment and technology have lead to increases in the number of islets that can be isolated from a single pancreas.

After successful isolation, the islets can be injected through a catheter into the patient's liver during a thirty-minute procedure. A group of doctors at the University of Alberta in Edmonton, Canada has had promising results in human islet transplantation. Normal sugar levels have been documented after human islet transplants. Also, recent improvements in immunosuppressive drug treatments have resulted in sustained insulin-independence in selected type 1 diabetic patients. The traditional method of transplant immunosuppression includes using some form of a steroid drug. Steroids have been found to injure or kill the islets after transplant. The doctors in Edmonton, Canada established an immunosuppression formula that does not use steroids. The objective of the study here at Emory University is to reproduce the successful results of human islet transplantation that have been achieved by the doctors at the University of Alberta using steroid free immunosuppression.

The Emory Islet Transplant Program will enroll ten patients, ages 18 to 65, in the study. Each of the ten patients will receive at least 2 islet transplants from 2 different organ donors. A third transplant may be required based on the patient's insulin requirements after the 1st two transplants. Each patient will be placed on immunosuppressive drugs to prevent the body from rejecting or destroying the transplanted islets. Each patient will have his/her blood sugar levels and insulin requirements monitored very closely after each transplant. The patients will also have various tests to determine if their diabetic complications improve, remain the same, or become worse. The patients will be asked to record any episodes of hypoglycemia or low blood sugars while participating in this study. Emory will examine whether or not there is a decrease in how often the episodes occur. Patients will also undergo regular eye exams to document retinal changes or improvements that may occur after transplant. At this time it is not known whether islet transplantation slows or stops the progression of common diabetic complications. More experience and research is needed before this can be determined. One focus of our research will be to study diabetic complications in patients who receive islet transplants.

The major goal of the Emory Islet Transplant Program is for patients participating in this study to be free of the need for insulin injections after 2 islet transplants. Because many advances have been made in islet transplantation, the transplant team at Emory would like to participate in this promising treatment of type 1 diabetes and, most importantly, help those who suffer from this disease become free from daily insulin injections and avoid the devastating complications that happen as a result of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus diagnosed > 5 years previously
* Body mass index less than or equal to 26
* 18 to 65 years of age
* Compliance with an optimized diabetic management plan as assessed by an Emory University endocrinologist
* Checking and recording blood sugars at least 3 times per day
* Intensive insulin therapy (injecting insulin at least 3 times a day or using an insulin pump)
* Severe hypoglycemia and/or hyperglycemia. Severe hypoglycemia is defined by: episodes requiring assistance by others and/or hypoglycemic unawareness (the inability to recognize blood glucose < 54 mg/dL). Severe hyperglycemia is defined by: two episodes of ketoacidosis requiring hospitalization within the past year.

Exclusion Criteria:

* Renal dysfunction
* Severe co-existing cardiac disease, characterized by any one of these conditions: recent myocardial infarction (within past six months); angiographic evidence of non-correctable coronary artery disease; or evidence of ischemia on a dobutamine stress echocardiogram.
* Current bacterial or fungal infection
* Macroproteinuria
* Baseline hemoglobin < 11.4 gm/dL in women; < 12.9 gm/dL in men.
* Hyperlipidemia
* Positive tests for human immunodeficiency virus (HIV), or hepatitis B or C
* Negative antibody test for varicella zoster virus (subjects may be reconsidered if they receive the vaccination and convert to a positive antibody)
* History of malignancy (except squamous or basal cell skin carcinoma)
* Previous/concurrent organ transplantation
* Presence of HLA panel reactive antibodies > 20%
* Active peptic ulcer disease
* Evidence of gallbladder disease including cholecystitis and cholelithiasis
* Evidence of liver disease including hepatic neoplasm, portal hypertension, or persistently abnormal liver function tests.
* Persistent coagulopathy or current use of anticoagulants (not including aspirin)
* Sickle cell anemia
* Positive pregnancy test, intent for future pregnancy, failure to follow effective contraceptive measures, or presently breastfeeding
* Active alcohol or substance abuse. This includes smoking (must be abstinent for six months). Active alcohol abuse should be considered using the current National Institute on Alcohol Abuse and Alcoholism (NIAAA) definitions.
* Psychiatric disorder making the subject not a suitable candidate for transplantation
* Current use of systemic steroid medications
* Evidence of insulin resistance (insulin requirement > 1.2 units/kg/day)
* Inability to provide informed consent
* Any condition or any circumstance that makes it unsafe to undergo an islet transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2002-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole A Turgeon, MD, Principal Investigator — Emory University; Christian P. Larsen, MD DPhil, Principal Investigator — Emory University
Locations (1):
- The Emory Transplant Center, Atlanta, Georgia, United States

REFERENCES:
- [Result] Turgeon NA, Avila JG, Cano JA, Hutchinson JJ, Badell IR, Page AJ, Adams AB, Sears MH, Bowen PH, Kirk AD, Pearson TC, Larsen CP. Experience with a novel efalizumab-based immunosuppressive regimen to facilitate single donor islet cell transplantation. Am J Transplant. 2010 Sep;10(9):2082-91. doi: 10.1111/j.1600-6143.2010.03212.x. PMID 20883542
- See also: Juvenile Diabetes Research Foundation, non-profit organization, sponsor of this study — http://www.jdrf.org
- See also: Emory Transplant Center website — http://transplant.emory.edu/index.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten participants fulfilled entry criteria and were listed for islet transplantation. Prior to receiving the transplant, one of the participants became ineligible while on the organ donor waiting list due to glucose control being stabilized with an insulin pump, and an additional participant was lost to follow up.
Period: Overall Study
Arm/Group | Islet Transplant
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants who received islet transplantation
Groups:
- Islet Transplant: 10 subjects were found eligible and were can be matched to an appropriate donor will receive/have received an islet transplant---1 INELIGIBLE WHILE ON WAITLIST.
  Transplantation of Human Islets: Human islets, at least 9,000 islet equivalents per kilogram of body weight. Transplant involves surgical procedure
Arm/Group | Islet Transplant
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Insulin-Independent Subjects at One Year Following Islet Cell Transplantation
Description: Independence from insulin injections is measured by the actual use of insulin by the study participants.
Time Frame: one year after transplant
Measure: Number; unit: participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 8
participants | 5

2. Secondary Outcome: Number of Insulin-independent Subjects Following Islet Transplantation
Description: Participants who did not need to take insulin at 1, 3, 6, 12, 18, 24, 36, 48 and 60 months following islet transplantation
Time Frame: 1, 3, 6, 9,12,18, 24, 36, 48 and 60 months post-transplantation
Measure: Number; unit: participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 8
participants
  1 Month Post-Transplant | 6
  3 Months Post-Transplant | 6
  6 Months Post-Transplant | 6
  9 Months Post-Transplant | 6
  12 Months Post-Transplant | 5
  18 Months Post-Transplant | 5
  24 Months Post-Transplant | 5
  36 Months Post-Transplant | 3
  48 Months Post-Transplant | 2
  60 Months Post-Transplant | 2

3. Secondary Outcome: Number of Subjects With HbA1C ≤ 6.5%
Description: HbA1C was assessed in subjects 1, 3, 6, 9,12,18,24, 36, 48 and 60 months after transplantation and the number of subjects with values ≤ 6.5% was recorded which indicated better control of blood glucose levels.
Time Frame: 1, 3, 6, 9,12,18,24, 36, 48 and 60 months post-transplantation
Measure: Number; unit: participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 8
participants
  1 Month Post-Transplant | 6
  3 Months Post-Transplant | 7
  6 Months Post-Transplant | 8
  9 Months Post-Transplant | 8
  12 Months Post-Transplant | 8
  18 Months Post-Transplant | 8
  24 Months Post-Transplant | 7
  36 Months Post-Transplant | 6
  48 Months Post-Transplant | 5
  60 Months Post-Transplant | 4

4. Secondary Outcome: The Number of Subjects Exhibiting Fasting C-peptide Levels ≥ 0.5 ng/mL
Description: Number of Participants With Endogenous Insulin Production Post-transplant, Assessed by Fasting C-peptide Levels at 1, 3, 6, 9,12,18, 24, 36, 48 and 60 months after islet cell transplantation
Time Frame: 1, 3, 6, 9,12,18, 24, 36, 48 and 60 months post-transplantation
Measure: Number; unit: participants
Arm/Group | Islet Transplant
Number analyzed (Participants) | 8
participants
  1 Month Post-Transplant | 6
  3 Months Post-Transplant | 6
  6 Months Post-Transplant | 6
  9 Months Post-Transplant | 6
  12 Months Post-Transplant | 5
  18 Months Post-Transplant | 5
  24 Months Post-Transplant | 5
  36 Months Post-Transplant | 5
  48 Months Post-Transplant | 3
  60 Months Post-Transplant | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for as long as the study participants were willing to be followed for safety monitoring. The follow up time ranged from 3 years to 5 years and 9 months.
Arm/Group | Islet Transplant
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplant (N=8)
Hospitalization for diarrhea, nausea, vomiting, and abdominal pain (Gastrointestinal disorders) | 1 (1) — Hospitalization for diarrhea, nausea, vomiting, and abdominal pain management
Pneumonia (Infections and infestations) | 1 (1) — Pneumonia with bilateral pleural effusions
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Islet Transplant (N=8)
Anemia (Blood and lymphatic system disorders) | 7
Diarrhea (Gastrointestinal disorders) | 7
Elevated Liver Enzymes (Hepatobiliary disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 8
Mouth Ulcers (Skin and subcutaneous tissue disorders) | 8
Abdominal Hernia (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes